CLINICAL TRIAL: NCT07088081
Title: Evaluation of Efficacy and Safety of Immune Check Point Inhibitors in Hepatocellular Carcinoma Patients in Ain Shams University Hospitals
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD111/2025
Record Dates: First submitted 2025-07-05; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: HCC - Hepatocellular Carcinoma; Immunotherapy; Immune Checkpoint Therapy; Immune Checkpoint Inhibitor-Induced Dermatitis; Atezolizumab and Bevacizumab in Hepatocellular Carcinoma; Durvalumab
Keywords: Immune check points inhibitors efficacy; Immune check points inhibitors safety; Response evaluation in hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the response to immunotherapy in HCC, assess the toxicity profile and measure overall survival within the study period. The primary end point is evaluation of progression free survival in HCC patients receiving immunotherapy. The secondary end point is to assess overall survival within the study period, duration of response and the response rate. The tertiary end point is to assess the toxicity profile.

DETAILED DESCRIPTION:
Treatment starts after MDT discussion and approval for diagnosis, staging and treatment protocol.

* This study includes patients with advanced HCC who will receive their first line of treatment. Cases will receive atezolizumab (1200 mg) + bevacizumab (15mg/kg) every 3 weeks or Tremilimumab (300 mg single dose IV infusion on first day only) + Durvalumab (1500 mg on the same day then every 4 weeks) according to eligibility criteria.
* Cases will be evaluated every cycle clinically and laboratory.
* Baseline investigations will include;

  1. Laboratory ;

     1. CBC
     2. liver enzymes (ALT, AST, alkaline phosphatase, GGT)
     3. liver function tests (serum albumin, serum bilirubin total and direct, INR)
     4. kidney function tests (serum creatinine, BUN, 24 hrs urinary protein)
     5. electrolytes Na, K, Ca)

     t) Others; HBAlc, Thyroid function tests (TSH, T3, T4), Alpha feto protein
  2. Radiological imagings;

     1. Triphasic CT and/or dynamic MRI abdomen
     2. PET scan or CT chest and bone scan
     3. ECG, ECHO, Upper GI endoscopy
* Every 3 months patients will undergo laboratory and radiological investigations, assessed by 2 blinded radiologists.
* The degree of adverse events was evaluated according to The Common Terminology Criteria for Adverse Events version 5.0.(30) ,which rates toxicity on a scale from 1 to 5, with ascending order of severity. This will be managed according to toxicity grade whether treatment interruption, dose reduction or discontinuation.
* Study treatment to be continued until disease progression, unacceptable toxicity, serious inter-current illness, patient request for discontinuation, or need for any other anticancer agent other than study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* Hepatocellular carcinoma based on histological diagnosis or the typical findings on radiological imaging including enhanced dynamic computed tomography (CT) and/or dynamic magnetic resonance imaging (MRI).
* ECOG Performance status of 0 or 1
* Patients with Child-Pugh class A
* BCLC stage B with diffuse, infiltrative, or extensive bilobar involvement
* BCLC stage B with tumor progression after failure of TACE
* BCLC stage C
* No prior systemic therapy for HCC
* Additional eligibility criteria; Hb ≥ 9 g/dl, platelets ≥ 75x10%/1, ANC ≥ 1.5 x10% for Atezolizumab/bevacizumab and ANC ≥ 1x10%1 for Durvalumab/Tremilimumab, INR ≤ 2, albumin ≥ 2.8 g/dl, total bilirubin

  ≤ 3 mg/dl, AST and ALT ≤ 5 x ULN, creatinine clearance ≥ 50 ml/min
* Additional criteria for Atezolizumab/Bevacizumab; upper endoscopy showing no risky high grade esophageal varices (within 6 months of first dose) unless adequately managed

Exclusion Criteria:

* Performance status ≥ 2
* Patients with Child-Pugh class B or C
* BCLC stage A or D
* Active tuberculosis or active human immunodeficiency virus (HIV) infection
* HCV or HBV infection except if; HBV DNA < 500 IU/ml or started anti- HBV treatment for a minimum of 14 days prior to first dose
* Severe infection requiring hospitalization within 4 weeks prior to first dose
* History of allogenic stem cell or solid organ transplant
* Treatment with systemic immunostimulatory or immunosuppressive medication
* Active and history of autoimmune disease or immune deficiency
* Receiving a live, attenuated vaccine within 4 weeks prior to first dose
* History of idiopathic pulmonary fibrosis, or evidence of active pneumonitis
* Central nervous system metastases
* Symptomatic hypercalcemia (ionized calcium > 1.5 mmol/1 (6 mg/dl), calcium > 12 mg/dl, or corrected serum calcium > ULN)
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Cardiac conditions, such as severe heart failure, unstable angina, recent myocardial infarction, severe arrhythmias
* Evidence of bleeding diathesis or coagulopathy Special for atezolizumab + bevacizumab
* Risky esophageal or gastric varies unless adequately managed
* Severe portal hypertensive gastropathy which is associated with decline in hemoglobin, uniess controlled
* Severe proteinuria ≥ 3.5 g/24 hrs or by dipstick 4+ proteinuria, according to CTCAE. Special for tremelimumab + durvalumab
* Main portal vein tumor thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling for patients fulfilling the eligibility criteria and after multidisciplinary team discussion at Clinical oncology department and HCC clinics, Ain Shams University Hospitals, Cairo.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival in HCC patients receiving immunotherapy. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival (PFS) is defined as the time elapsed between treatment initiation and tumor progression or death from any cause. Progression (i.e., PD) was defined as presence of new measurable/non- measurable lesions, or ≥ 20% increase in tumour burden relative to nadir

SECONDARY OUTCOMES:
overall survival within the study period, | From date of randomization until the date of loss of follow up or date of death from any cause, whichever came first, assessed up to 12 months
  Overall survival (OS) is defined as time from diagnosis to either last follow-up or /death
Response rate | From enrollment to study till 1 year or treatment
  Response rate is defined as the proportion of patients with a complete response/immune complete response or partial response/ immune partial response to treatment

OTHER OUTCOMES:
Assess the toxicity profile of immunotherapy | From enrollment to 1 year of treatment
  The degree of adverse events was evaluated according to The Common Terminology Criteria for Adverse Events version 5.0. ,which rates toxicity on a scale from 1 to 5, with ascending order of severity. This will be managed according to toxicity grade whether treatment interruption, dose reduction or discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasya, Egypt